CLINICAL TRIAL: NCT00419276
Title: Effect of Ambulatory Continuous Femoral Nerve Blocks on Readiness-for-Discharge Following Total Knee Arthroplasty: A Multicenter, Randomized, Triple-Masked, Placebo-Controlled Investigation
Brief Title: Effect of Ambulatory Continuous Femoral Nerve Blocks on Readiness-for-Discharge Following Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University of Florida (Other); Stryker Instruments (Industry)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, in Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PAINfRE TKA Investigation; 1K23GM077026-01A1 (NIH)
Record Dates: First submitted 2007-01-04; First posted 2007-01-08 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Total Knee Arthroplasty
Keywords: Total knee arthroplasty, postoperative analgesia; Primary, unilateral, total knee arthroplasty

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prolonged infusion (Experimental): At least 100 hours of femoral perineural ropivacaine infusion.
  Interventions: Procedure: Ambulatory continuous femoral nerve block for 100 hours
- Standard-of-Care (Placebo Comparator): Overnight femoral perineural ropivacaine infusion followed by a femoral perineural normal saline infusion (placebo) until postoperative day 4.
  Interventions: Procedure: Ambulatory continuous femoral nerve block for 100 hours

INTERVENTIONS:
Procedure: Ambulatory continuous femoral nerve block for 100 hours — Treatment group: 100 hours of ropivacaine femoral perineural infusion. Standard-of-care group: overnight ropivacaine femoral perineural infusion followed by a normal saline infusion.

SUMMARY:
To determine if following total knee replacement, putting local anesthetic-or numbing medication-for five days through a tiny tube next to the nerves that go to the knee will decrease the time that patients need to spend in the hospital.

DETAILED DESCRIPTION:
1. Procedures that will be done as part of your normal clinical care (even if you do not participate in this research):

   You will have some monitors placed (such as a blood-pressure cuff) and be given some medicines through your intravenous line to make you very sleepy. The anesthesiologist will then place a tiny tube, called a catheter, near your nerves that will be used during and following surgery. This involves carefully cleaning the immediate area in the upper thigh where the catheter will be placed, numbing the site of the catheter with local anesthetic placed just under the skin, placing a needle through the skin that is numbed to an area near where your nerves are, putting the catheter through the needle so that the tip is next to your nerves, then removing the needle leaving the catheter in place. You can still go to sleep for the surgery, but you will be more comfortable when you wake up because the numbing medicine will be working to take away much of the pain. If you are not part of this study, you would go from the recovery room to a room in the hospital for 3-5 days, and your catheter would probably be removed the morning after surgery. After removal of your catheter, you would depend on oral and intravenous pain medicine ("opioids"-like morphine) to control your surgical pain. You would go home with only oral opioids since intravenous opioids cannot be provided at home.
2. Procedures that will be done only if you participate in this research study:

   From the recovery room you will go to the surgical ward. During your stay in the hospital you will have the ability to push a button on a small infusion pump-a little device that holds and puts the medicine through the catheter to bath your nerves in local anesthetic-to give yourself more medicine through the tube to your nerves if you have pain. If this does not help enough, you will take pain pills to help. And if this does not help enough, you will be given opioids (strong pain medicine like morphine) into your intravenous line.
3. On the morning after surgery, the medicine in your little infusion pump will be replaced by either (1) more medicine, or (2) salt water, or "normal saline". The pharmacist will determine this randomly-like flipping a coin-and neither you nor the doctors/nurses caring for you will know which you have. This is to keep any of us from inadvertently/ unconsciously affecting the results of the study.
4. You will undergo physical therapy and following this you will be checked to see if you are ready to go home. This will include walking in the morning and afternoon with a physical therapist. When you are ready to go home beginning on the third day after surgery, you may go home with the little infusion pump and the tube that delivers the fluid. You will be given a prescription for pain pills in case you need them for pain relief.
5. One of the study investigators will call you each night to ensure that you are comfortable for the first 6 nights after your surgery, and you will be given the phone and pager numbers of your physician (anesthesiologist) available for you to contact 24 hours/day, 7 days/week. A research nurse will call you for five nights beginning the day after surgery to ask about your comfort level and other study-related information such as your satisfaction level.
6. On the fourth evening following surgery your catheter will be removed. You have two options available to you to remove your catheter. You can call a physician who will talk you or your caregiver through this process over the phone--it will not hurt or bleed. Your other option is to come back to the hospital to have a health care professional remove the catheter for you. The pump, catheter and remaining fluid are disposable and will not hurt people or pets, so they will be thrown away. A physician will call you the night after the catheter comes out to ensure that you are comfortable.
7. A research nurse will call you at 7 days and then 1, 2, 3, 6, and 12 months following your surgery. Each of these calls will be less than five minutes in length during which time you will be asked questions about your levels of pain, stiffness and joint functional ability. Your participation will be limited to 12 months after surgery with these phone calls.

ELIGIBILITY:
Inclusion Criteria:

1. undergoing primary, unilateral knee replacement
2. age 18 - 75 years
3. postoperative analgesic plan includes perineural local anesthetic infusion and
4. the availability of a "caretaker" who will remain with the patient from home discharge until catheter removal.

Exclusion Criteria:

1. morbid obesity as defined by a body mass index > 40 (BMI=weight in kg / [height in meters]2)
2. renal insufficiency (preoperative creatinine > 1.5 mg/dL)
3. chronic opioid use (use within the 2 weeks prior to surgery and duration of use > 4 weeks)
4. history of opioid abuse and
5. any comorbidity which results in moderate or severe functional limitation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2007-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The time from surgical stop until patients meet three readiness-for-discharge criteria (adequate analgesia, free of intravenous opioids for 12 hours, able to ambulate at least 30 meters). | Twice daily until hospital discharge

SECONDARY OUTCOMES:
Quality-of-life as measured with the Western Ontario McMasters University questionnaire (WOMAC) up to 1 year postoperatively. | preoperatively, then 7 days, 1, 2, 3, 6, and 12 months postoperatively
In addition, we will evaluate daily pain scores; (2) daily oral and intravenous opioid requirements; (3) sleep quality and disturbances; (4) knee flexion and extension; and (5) patient satisfaction. | Daily until 6 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, MD, MS, Principal Investigator — University of California, San Diego
Locations (4):
- United States (3):
  - Alta Bates Summit Medical Center, Berkeley, California
  - University of California San Diego, San Diego, California
  - University of Florida, Gainesville, Florida
- Sunnybrook Health Sciences Centre and the Holland Orthopedic and Arthritic Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Ilfeld BM, Gearen PF, Enneking FK, Berry LF, Spadoni EH, George SZ, Vandenborne K. Total knee arthroplasty as an overnight-stay procedure using continuous femoral nerve blocks at home: a prospective feasibility study. Anesth Analg. 2006 Jan;102(1):87-90. doi: 10.1213/01.ane.0000189562.86969.9f. PMID 16368810
- [Derived] Ilfeld BM, Shuster JJ, Theriaque DW, Mariano ER, Girard PJ, Loland VJ, Meyer S, Donovan JF, Pugh GA, Le LT, Sessler DI, Ball ST. Long-term pain, stiffness, and functional disability after total knee arthroplasty with and without an extended ambulatory continuous femoral nerve block: a prospective, 1-year follow-up of a multicenter, randomized, triple-masked, placebo-controlled trial. Reg Anesth Pain Med. 2011 Mar-Apr;36(2):116-20. doi: 10.1097/aap.0b013e3182052505. PMID 21425510
- See also: PAINfRE multicenter study research investigators — http://www.painfre.com